CLINICAL TRIAL: NCT06354309
Title: Impact of Different Types of Virtual Reality Games on Motion Sickness and Ocular in Adults: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: He Eye Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: VR_Study
Record Dates: First submitted 2024-04-03; First posted 2024-04-09 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Amblyopia; Motion Sickness; Dry Eye
Keywords: Visual function training; Amblyopia; Virtual reality; Motion Sickness; Dry eye
MeSH Terms: conditions — Amblyopia; Motion Sickness; Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pre and post control study (Experimental): The subjects used the HMVR for 2 sessions of game training (30 minutes each, 10 minutes intervals).
  Interventions: Other: Virtual reality game

INTERVENTIONS:
Other: Virtual reality game — Pre and post control study after use virtual reality game

SUMMARY:
The research project titled "The Impact of Immersive Virtual Reality Training on Adult: Motion Sickness, and Ocular Surface: A Pilot Study" aimed to evaluate the initial safety impact of head-mounted virtual reality (HMVR) devices with virtual reality amblyopia training games on postural stability, motion sickness, and ocular surface in healthy adult participants. 38 adults (76 eyes) with normal corrected vision and stereo vision were recruited. All subjects used HMVR device for two consecutive training sessions (30 minutes each, 10 minutes intervals). Before training, after the first training and the second training, recorded the results including best corrected visual acuity (BCVA), ocular position, stereo vision, postural stability, non-invasive tear breakup time (NITBUT), tear meniscus height (TMH), red eye analysis, lipid layer classification (TFLL), eye blink frequency, eye surface temperature, simulator sickness questionnaire (SSQ) score, ocular surface disease index (OSDI) dry eye questionnaire score, visual quality questionnaire score and visual fatigue questionnaire score.

DETAILED DESCRIPTION:
1. Title: The Impact of Immersive Virtual Reality Training on Adult: Motion Sickness, and Ocular Surface: A Pilot Study.
2. Purpose: To evaluate the initial safety impact of head-mounted virtual reality (HMVR) devices with virtual reality amblyopia training games on postural stability, motion sickness, and ocular surface in healthy adult participants.
3. Methods: A total of 38 healthy adult volunteers (18 males, 20 females) aged 18-42 years old were recruited from Shenyang He Eye Specialist Hospital from July to August 2023. Inclusion criteria: age ≥18 years; BCVA >=1.0; Titmus is between 40-60 ". Exclusion criteria: history of eye surgery and trauma within 3 months; Active eye problems; Pregnancy or lactation; Those who were determined by the investigator to be unsuitable for this study. This study was approved by the Ethics Committee of Shenyang He Eye Specialist Hospital (IRB(2023)K023.01).

3.1Research equipment Pico VR all-in-one (Neo2 Lite, Hainan Creative Vision Future Technology Co., LTD., China (referred to as "PICO") is a VR headset, which is used together with BeiShiYou visual function training software (BV-2, Shenyang BeiYou Technology Co., LTD., referred to as "BeiShiYou") 3.2 Procedure The procedure was divided into four steps: A. Sign the informed consent. B. First ophthalmic examination (diopter, BCVA, ocular position, stereo vision, postural stability, non-invasive tear breakup time, tear meniscus height, red eye analysis, lipid layer classification, eye blink frequency, eye surface temperature) and questionnaires survey (simulator sickness questionnaire, semans balance disorder scale, ocular surface disease index dry eye questionnaire, visual quality questionnaire and visual fatigue questionnaire). C. Conduct the first VR headset game training for 30 minutes, and then conduct the second eye examination and questionnaire survey above. D. Conduct the second VR headset game training for 30 minutes, and then conduct the third eye examination and questionnaire survey above (Figure 2).

3.3 Observation Indicators includes Simulator sickness questionnaire (SSQ), Postural stability, Non-invasive tear breakup time (NITBUT), Tear meniscus height, Lipid layer classification, Eye blink frequency, Central ocular surface temperature, Dry eye questionnaire score, Visual quality questionnaire score, Visual fatigue score.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18
* Best vision >=1.0
* Titmus is between 40s and 60s

Exclusion Criteria:

* History of eye surgery and trauma within 3 months
* Active eye diseases
* Pregnancy and lactation period
* Allergic to fluorescein sodium
* The researcher determined that the subjects were not suitable for this study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-10-20 (Actual)

PRIMARY OUTCOMES:
Simulator Sickness Questionnaire Score | Baseline, 30min, 60min
  Record the simulator sickness questionnaire score after use virtual reality game

SECONDARY OUTCOMES:
Postural stability | Baseline, 30min, 60min
  Record the postural stability level after use virtual reality game
Non-invasive tear breakup time | Baseline, 30min, 60min
  Check with Eye Surface Analyzer (OCULUS, Germany)
Tear meniscus height | Baseline, 30min, 60min
  Check with Eye Surface Analyzer (OCULUS, Germany)
Lipid layer classification | Baseline, 30min, 60min
  Check with DR-1 dry eye measurement
Eye blink frequency | Baseline, 30min, 60min
  Collect the blink frequency with DJI Pocket 2 Creator Combo (Shenzhen DJI Innovation Technology Co., LTD.)
Eye surface temperature | Baseline, 30min, 60min
  Collect eye surface temperature with Flir ONE Pro mobile phone Infrared thermal camera for Apple IOS (Teledyne FLIR, USA)
Ocular surface disease index dry eye questionnaire score | Baseline, 30min, 60min
  Record with OSDI questionaire
Visual quality questionnaire score | Baseline, 30min, 60min
  Record with visual quality questionnaire
Visual fatigue questionnaire score | Baseline, 30min, 60min
  Record with visual fatigue questionaire

CONTACTS AND LOCATIONS:
Overall Officials: Ling Xu, MD, Principal Investigator — He Eye Hospital
Locations (1):
- He Eye Hospital, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No